CLINICAL TRIAL: NCT05631717
Title: A Prospective, Single-center Study of Comparing the Efficacy and Safety of Human Umbilical Cord Mesenchymal Stem Cells and Low-dose IL-2 in the Treatment of Lupus Nephritis
Brief Title: The Study of Comparing the Efficacy and Safety of Human Umbilical Cord MSCs and Low-dose IL-2 in the Treatment of LN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-LCYJ-MS-38
Record Dates: First submitted 2022-11-13; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-09

CONDITIONS: Systemic Lupus Erythematosus; Lupus Nephritis
Keywords: Mesenchymal stem cells; interleukin-2
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis | interventions — Interleukin-2; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Intervention Model Description: The test will be divided into two groups. One group of subjects will receive intravenous injection of human umbilical cord mesenchymal stem cells (2 × 106 cells/kg body weight, suspended in 30ml of normal saline); the other group will receive IL-2 (1 × 106 IU) every other day. Subcutaneous injection for 2 weeks (a total of 7 injections), with an interval of 2 weeks, such that 4 weeks is a cycle, and three consecutive cycles of treatment for a total of 12 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSCs group (Experimental): In this group, patients will receive intravenous injection of human umbilical cord mesenchymal stem cells (2 × 10^6 cells / kg body weight, suspended in 30ml saline)
  Interventions: Biological: Human umbilical cord mesenchymal stem cells
- IL-2 group (Experimental): In this group, patients will receive subcutaneous injection of IL-2 (1×10^6IU) every other day for 2 weeks (7 times), with an interval of 2 weeks.
  Interventions: Drug: Interleukin-2

INTERVENTIONS:
Biological: Human umbilical cord mesenchymal stem cells — Human umbilical cord mesenchymal stem cells (1 × 10 ^6 cells / kg body weight, suspended in 30ml saline), intravenous drip once.
  Arms: MSCs group
Drug: Interleukin-2 — IL-2 (1×10^6IU) will be injected subcutaneously every other day for 2 weeks (7 times), with an interval of 2 weeks. 4 weeks is a cycle, and three cycles were continuously treated for 12 weeks.
  Other Names: Recombinant Human Interleukin-2(1) for Injection
  Arms: IL-2 group

SUMMARY:
The purpose of this study is to compare the efficacy and safety of human umbilical cord mesenchymal stem cells and low-dose IL-2 in the treatment of LN

DETAILED DESCRIPTION:
Allogeneic MSC transplantation has shown significant efficacy and good safety in the treatment of refractory autoimmune diseases such as lupus nephritis (LN), and has a broad application prospect. One of its mechanisms is that MSCs up-regulates the production of IL-2 and promotes the production of Treg cells. The breakthrough in this technology has brought new hope for patients with autoimmune diseases. Some small sample studies at home and abroad have shown that low-dose IL-2 can be used to treat LN. Recently, the research team found that a single dose of IL-2 showed a longer effect than repeated low-dose MSCs. However, there is still a lack of prospective randomized studies to confirm that the efficacy of allogeneic MSC is better than that of low-dose IL-2. Therefore, carrying out this prospective randomized study will make a real breakthrough in the clinical application of MSC in SLE, and open up a new field for the treatment of SLE for the benefit of mankind.

ELIGIBILITY:
Inclusion Criteria:

Only patients with active lupus nephritis who meet all of the following criteria are eligible for inclusion in this study:

* Before random assignment, records show that it meets at least 4 of the 11 SLE classification criteria recommended by ACR in 1997.
* Age: age > 18 years old, ≤ 65 years old when obtaining informed consent
* SLEDAI-2K score ≥ 6
* Urinary total protein / creatinine ratio > 1.0 or 24-hour urinary protein > 1.0g, with or without microscopic hematuria
* If they are fertile, they must agree to use effective contraception during the trial.
* In the case of women of childbearing age, urinary pregnancy and serum pregnancy tests should be negative.
* Voluntarily sign informed consent and comply with the requirements of the research programme

Exclusion Criteria:

Patients who met any of the following criteria could not be enrolled in this study:

* Patients who had received rituximab or any other B cell depletion therapy within 24 weeks before screening; patients who received unstable doses of mycophenolate mofetil, cyclophosphamide or other immunosuppressants (including Cyclosporine, Tacrolimus, Tripterygium wilfordii, Leflunomide, Azathioprine, Iguratimod) within the first 12 weeks of screening. Received biological agents or small molecule targeted drugs for immune diseases within 4 weeks before screening, such as Etanercept, Infliximab, Adalimumab Solution, Golimumab, Belimumab, Tocilizumab or JAK inhibitors;
* Plasmapheresis or immunosorbent therapy within 12 weeks before screening.
* Accompanied by severe and uncontrolled cardiovascular diseases, nervous system diseases, lung diseases, liver diseases, endocrine and gastrointestinal diseases.
* Current or recent (within 4 weeks before random allocation) a history of severe active or recurrent bacterial, viral, fungal, parasitic or other infections (including, but not limited to, tuberculosis and atypical mycobacterial diseases, hepatitis B and C, HIV infection, herpes zoster, but excluding onychomycosis). Or any infected person who needs hospitalization and intravenous antibiotic treatment within 4 weeks before screening or any infected person who needs treatment within 2 weeks before screening.
* Any major surgery has been performed within 12 weeks before screening, or major surgery is required during the study period, which the researchers believe will pose an unacceptable risk to the patient;
* Live vaccine will be given within 12 weeks before random allocation, or live vaccine is expected to be needed / received during the study (except for herpes zoster vaccination).
* Patients with a history of malignant tumors, including solid tumors and hematological malignancies (except for excised or cured basal cell carcinoma of the skin);
* Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Response rates in both groups （CR and RR） | 24 Weeks
  Complete response (CR): serum creatinine ≤ 1.2 mg/dl or ≤125% of baseline, and ratio of protein in morning urine to creatinine <0.5 or 24-hour urine protein quantification < 0.5 g, and prednisone reduced to ≤10 mg/day (or equivalent).
  Partial response (PR): if serum creatinine and ratio of protein in morning urine to creatinine (or 24-hour urine protein quantification) were abnormal before treatment, both improved by >30% after treatment, and there were no other indicators of deterioration; If only the ratio of protein in morning urine to creatinine (or 24-hour urine protein quantification) is abnormal before treatment, the improvement is >50% after treatment.

SECONDARY OUTCOMES:
Time for both groups of subjects to achieve PR and CR | 24 Weeks
  Complete response (CR): serum creatinine ≤ 1.2 mg/dl or ≤125% of baseline, and ratio of protein in morning urine to creatinine <0.5 or 24-hour urine protein quantification < 0.5 g, and prednisone reduced to ≤10 mg/day (or equivalent).
  Partial response (PR): if serum creatinine and ratio of protein in morning urine to creatinine (or 24-hour urine protein quantification) were abnormal before treatment, both improved by >30% after treatment, and there were no other indicators of deterioration; If only the ratio of protein in morning urine to creatinine (or 24-hour urine protein quantification) is abnormal before treatment, the improvement is >50% after treatment.
SRI response status | 24 Weeks
  SRI response status at Week 24 Clinical efficacy will be measured using the SLE Responder Index (SRI), a composite endpoint that incorporates SLEDAI-2K, BILAG 2004, and a visual analog scale (VAS) of physician-rated disease activity to determine patient improvement.
SLEDAI-2K score and change from baseline | Baseline, Week 4, 8, 16, 20 and 24
  To describe the effect of treatment with MSCs or IL-2 using patient reported outcomes
BILAG-2004 score and change from baseline | Baseline, Week 4, 8, 16, 20 and 24
  To describe the effect of treatment with MSCs or IL-2 using patient reported outcomes
Hormone dosage and change from baseline | Baseline, Week 4, 8, 16, 20 and 24
  To describe the effect of treatment with MSCs or IL-2 using dose of hormones in patients
Patient incidence of Treatment-Emergent Adverse Events | 24 Weeks
  To characterize the safety of MSCs and IL-2
Patient incidence of Serious adverse events | 24 Weeks
  To characterize the safety of MSCs and IL-2
Number of patients with significant changes in laboratory values | 24 Weeks
  To characterize the safety of MSCs and IL-2
Number of patients with significant changes in vital signs | 24 Weeks
  To characterize the safety of MSCs and IL-2

CONTACTS AND LOCATIONS:
Overall Officials: Jun Liang, Doctor, Study Chair — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School; Huayong Zhang, Doctor, Study Director — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School; Cheng Zhao, Doctor, Study Director — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School; Linyu Geng, Doctor, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School; Xue Xu, Doctor, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School; Xiaolei Ma, Doctor, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School; Lihui Wen, Doctor, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School; Saisai Huang, Doctor, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School; Yunxia Yan, Master, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Geng L, Xu X, Zhang H, Chen C, Hou Y, Yao G, Wang S, Wang D, Feng X, Sun L, Liang J. Comprehensive expression profile of long non-coding RNAs in Peripheral blood mononuclear cells from patients with neuropsychiatric systemic lupus erythematosus. Ann Transl Med. 2020 Mar;8(6):349. doi: 10.21037/atm.2020.03.25. PMID 32355793
- [Background] Liang J, Zhang H, Kong W, Deng W, Wang D, Feng X, Zhao C, Hua B, Wang H, Sun L. Safety analysis in patients with autoimmune disease receiving allogeneic mesenchymal stem cells infusion: a long-term retrospective study. Stem Cell Res Ther. 2018 Nov 14;9(1):312. doi: 10.1186/s13287-018-1053-4. PMID 30428931
- [Background] Zhang H, Liang J, Qiu J, Wang F, Sun L. Ultrasonographic evaluation of enthesitis in patients with ankylosing spondylitis. J Biomed Res. 2017 Jan 19;31(2):162-169. doi: 10.7555/JBR.31.20160088. PMID 28808198
- [Background] Zhang H, Liang J, Tang X, Wang D, Feng X, Wang F, Hua B, Wang H, Sun L. Sustained benefit from combined plasmapheresis and allogeneic mesenchymal stem cells transplantation therapy in systemic sclerosis. Arthritis Res Ther. 2017 Jul 19;19(1):165. doi: 10.1186/s13075-017-1373-2. PMID 28724445
- [Background] Liang J, Zhang H, Zhao C, Wang D, Ma X, Zhao S, Wang S, Niu L, Sun L. Effects of allogeneic mesenchymal stem cell transplantation in the treatment of liver cirrhosis caused by autoimmune diseases. Int J Rheum Dis. 2017 Sep;20(9):1219-1226. doi: 10.1111/1756-185X.13015. Epub 2017 Feb 20. PMID 28217916
- [Background] Chen C, Liang J, Yao G, Chen H, Shi B, Zhang Z, Zhao C, Zhang H, Sun L. Mesenchymal stem cells upregulate Treg cells via sHLA-G in SLE patients. Int Immunopharmacol. 2017 Mar;44:234-241. doi: 10.1016/j.intimp.2017.01.024. Epub 2017 Jan 25. PMID 28129605
- [Background] Liang J, Wang F, Wang D, Zhang H, Zhao C, Wang S, Sun L. Transplantation of mesenchymal stem cells in a laryngeal carcinoma patient with radiation myelitis. Stem Cell Res Ther. 2015 Nov 4;6:213. doi: 10.1186/s13287-015-0203-1. PMID 26537898
- [Background] Liang J, Sun L. Mesenchymal stem cells transplantation for systemic lupus erythematosus. Int J Rheum Dis. 2015 Feb;18(2):164-71. doi: 10.1111/1756-185X.12531. Epub 2015 Jan 22. PMID 25611801
- [Background] Liang J, Zhang H, Wang D, Feng X, Wang H, Hua B, Liu B, Sun L. Allogeneic mesenchymal stem cell transplantation in seven patients with refractory inflammatory bowel disease. Gut. 2012 Mar;61(3):468-9. doi: 10.1136/gutjnl-2011-300083. Epub 2011 May 26. No abstract available. PMID 21617158
- [Background] Liang J, Li X, Zhang H, Wang D, Feng X, Wang H, Hua B, Liu B, Sun L. Allogeneic mesenchymal stem cells transplantation in patients with refractory RA. Clin Rheumatol. 2012 Jan;31(1):157-61. doi: 10.1007/s10067-011-1816-0. Epub 2011 Aug 12. PMID 21837432
- [Background] Liang J, Zhang H, Hua B, Wang H, Lu L, Shi S, Hou Y, Zeng X, Gilkeson GS, Sun L. Allogenic mesenchymal stem cells transplantation in refractory systemic lupus erythematosus: a pilot clinical study. Ann Rheum Dis. 2010 Aug;69(8):1423-9. doi: 10.1136/ard.2009.123463. PMID 20650877
- [Background] Liang J, Gu F, Wang H, Hua B, Hou Y, Shi S, Lu L, Sun L. Mesenchymal stem cell transplantation for diffuse alveolar hemorrhage in SLE. Nat Rev Rheumatol. 2010 Aug;6(8):486-9. doi: 10.1038/nrrheum.2010.80. Epub 2010 Jun 1. PMID 20517294